CLINICAL TRIAL: NCT03981796
Title: A Phase 3, Randomized, Double-blind, Multicenter Study of Dostarlimab (TSR-042) Plus Carboplatin-paclitaxel Versus Placebo Plus Carboplatin-paclitaxel in Patients With Recurrent or Primary Advanced Endometrial Cancer (RUBY)
Brief Title: A Study to Evaluate Dostarlimab Plus Carboplatin-paclitaxel Versus Placebo Plus Carboplatin-paclitaxel in Participants With Recurrent or Primary Advanced Endometrial Cancer
Acronym: RUBY
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Tesaro, Inc. (Industry)
Collaborators: European Network of Gynaecological Oncological Trial Groups (ENGOT) (Other); GOG Foundation (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 213361; ENGOT-EN6 (Other: ENGOT); GOG-3031 (Other: GOG); 4010-03-001 (Other: Tesaro); 2023-506551-23-00 (EU CTIS Number)
Record Dates: First submitted 2019-05-31; First posted 2019-06-11 (Actual); Last update posted 2025-09-03 (Actual); Status verified 2025-09

CONDITIONS: Neoplasms
Keywords: Dostarlimab; Carboplatin; Paclitaxel; Niraparib; Recurrent or primary advanced endometrial cancer; TSR-042
MeSH Terms: conditions — Neoplasms; Recurrence | interventions — dostarlimab; Carboplatin; Paclitaxel; niraparib

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The participant, Investigator, study staff, and the Sponsor study team and its representatives will be blinded to the assigned treatment.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Arm 1: Participants receiving dostarlimab + Carboplatin-paclitaxel followed by dostarlimab (Active Comparator)
  Interventions: Biological: Dostarlimab; Drug: Carboplatin; Drug: Paclitaxel
- Arm 2: Participants receiving placebo + carboplatin-paclitaxel followed by placebo (Placebo Comparator)
  Interventions: Drug: Placebo matching dostarlimab; Drug: Carboplatin; Drug: Paclitaxel
- Arm 3: Participants receiving dostarlimab + carboplatin-paclitaxel followed by dostarlimab+niraparib (Active Comparator)
  Interventions: Biological: Dostarlimab; Drug: Carboplatin; Drug: Paclitaxel; Drug: Niraparib
- Arm 4: Participants receiving placebo + carboplatin-paclitaxel followed by placebo (Placebo Comparator)
  Interventions: Drug: Placebo matching dostarlimab; Drug: Carboplatin; Drug: Paclitaxel; Drug: Placebo matching Niraparib

INTERVENTIONS:
Biological: Dostarlimab — Participants will be administered dostarlimab
  Other Names: TSR-042
  Arms: Arm 1: Participants receiving dostarlimab + Carboplatin-paclitaxel followed by dostarlimab; Arm 3: Participants receiving dostarlimab + carboplatin-paclitaxel followed by dostarlimab+niraparib
Drug: Placebo matching dostarlimab — Participants will be administered placebo matching dostarlimab
  Arms: Arm 2: Participants receiving placebo + carboplatin-paclitaxel followed by placebo; Arm 4: Participants receiving placebo + carboplatin-paclitaxel followed by placebo
Drug: Carboplatin — Participants will be administered carboplatin
Drug: Paclitaxel — Participants will be administered paclitaxel
Drug: Niraparib — Participants will be administered niraparib
  Arms: Arm 3: Participants receiving dostarlimab + carboplatin-paclitaxel followed by dostarlimab+niraparib
Drug: Placebo matching Niraparib — Participants will be administered placebo matching Niraparib
  Arms: Arm 4: Participants receiving placebo + carboplatin-paclitaxel followed by placebo

SUMMARY:
This is a 2 part study. Part 1 is to evaluate the efficacy and safety of dostarlimab plus carboplatin-paclitaxel followed by dostarlimab versus placebo plus carboplatin-paclitaxel followed by placebo; and Part 2 is to evaluate the efficacy and safety of dostarlimab plus carboplatin-paclitaxel followed by dostarlimab plus niraparib versus placebo plus carboplatin-paclitaxel followed by placebo in participants with recurrent or primary advanced (Stage III or IV) endometrial cancer.

ELIGIBILITY:
Inclusion Criteria:

Part 1 and Part 2:

* Female participant is at least 18 years of age.
* Participant has histologically or cytologically proven endometrial cancer with recurrent or advanced disease.
* Participant must have primary Stage III or Stage IV disease or first recurrent endometrial cancer with a low potential for cure by radiation therapy or surgery alone or in combination and meet at least one of the following criteria;

  1. Participant has primary Stage IIIA to IIIC1 disease with presence of evaluable or measurable disease per Response Evaluation Criteria in Solid Tumors (RECIST) version (v).1.1 based on Investigator's assessment. Lesions that are equivocal or can be representative of post-operative change should be biopsied and confirmed for the presence of tumor;
  2. Participant has primary Stage IIIC1 disease with carcinosarcoma, clear cell, serous, or mixed histology (containing greater than or equal to [>=] 10 percent carcinosarcoma, clear cell, or serous histology) regardless of presence of evaluable or measurable disease on imaging;
  3. Participant has primary Stage IIIC2 or Stage IV disease regardless of the presence of evaluable or measurable disease;
  4. Participant has first recurrent disease and is naïve to systemic anticancer therapy;
  5. Participant has received prior neo-adjuvant/adjuvant systemic anticancer therapy and had a recurrence or progression of disease (PD) >=6 months after completing treatment (first recurrence only).
* Participant has an ECOG performance status of 0 or 1.
* Participant has adequate organ function.

Part 2 only:

* Participants must have normal blood pressure (BP) or adequately treated and controlled hypertension (systolic BP lesser than or equal to [<=] 140 millimeter of mercury [mmHg] and diastolic BP <=90 mmHg).
* Participants must be able to take medication orally, by mouth (PO).

Exclusion Criteria:

Part 1 and Part 2:

* Participant has received neo-adjuvant/adjuvant systemic anticancer therapy for primary Stage III or IV disease and:

  1. has not had a recurrence or PD prior to first dose on the study OR
  2. has had a recurrence or PD within 6 months of completing systemic anticancer therapy treatment prior to first dose on the study.
* Participant has had >1 recurrence of endometrial cancer.
* Participant has received prior therapy with an anti-programmed cell death protein 1 (anti-PD-1), anti-PD-ligand 1 (anti-PD-L1), or anti-PD-ligand 2 (anti-PD-L2) agent.
* Participant has received prior anticancer therapy (chemotherapy, targeted therapies, hormonal therapy, radiotherapy, or immunotherapy) within 21 days or <5 times the half-life of the most recent therapy prior to Study Day 1, whichever is shorter.
* Participant has a concomitant malignancy, or participant has a prior non-endometrial invasive malignancy who has been disease-free for <3 years or who received any active treatment in the last 3 years for that malignancy. Non-melanoma skin cancer is allowed.
* Participant has known uncontrolled central nervous system metastases, carcinomatosis meningitis, or both.
* Participant has not recovered (that is [i.e.], to Grade <=1 or to Baseline) from cytotoxic therapy induced AEs or has received transfusion of blood products (including platelets or red blood cells) or administration of colony-stimulating factors (including granulocyte colony-stimulating factor [G-CSF], granulocyte macrophage colony-stimulating factor [GM-CSF], or recombinant erythropoietin) within 21 days prior to the first dose of study drug.
* Participant has not recovered adequately from AEs or complications from any major surgery prior to starting therapy.
* Participant is currently participating and receiving study treatment or has participated in a study of an investigational agent and received study treatment or used an investigational device within 4 weeks of the first dose of treatment.
* Participant is considered a poor medical risk due to a serious, uncontrolled medical disorder, nonmalignant systemic disease, or active infection requiring systemic therapy.
* Participant has received, or is scheduled to receive, a live vaccine within 30 days before first dose of study treatment, during study treatment, and for up to 180 days after receiving the last dose of study treatment.

Part 2 only:

* Participant has received prior therapy with a poly (adenosine diphosphate [ADP]-ribose) polymerase (PARP) inhibitor.
* Participant has clinically significant cardiovascular disease.
* Participant has any known history or current diagnosis of myelodysplastic syndrome (MDS) or acute myeloid leukemia (AML).
* Participant is at increased bleeding risk due to concurrent conditions.
* Participant has participated in Part 1 of this study

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 785 (Actual)
Dates: Start 2019-07-18 (Actual); Primary Completion 2026-11-26 (Estimated); Study Completion 2026-11-26 (Estimated)

PRIMARY OUTCOMES:
Parts 1 and 2: Progression-Free Survival (PFS) - investigator assessment | Up to 6 years
Part 1: Overall survival | Up to 6 years

SECONDARY OUTCOMES:
Part 2: Overall survival | Up to 6 years
Parts 1 and 2: Progression free survival (PFS) blinded independent central review (BICR) | Up to 6 years
Parts 1 and 2: Objective response rate (ORR) - BICR and Investigator assessment | Up to 6 years
Parts 1 and 2: Duration of response (DOR) - BICR and Investigator assessment | Up to 6 years
Parts 1 and 2: Disease control rate (DCR) - BICR and Investigator assessment | Up to 6 years
Parts 1 and 2: Patient-reported outcomes (PROs) in the European Quality of Life scale, 5-Dimensions, 5-Levels (EQ-5D-5L) | Up to 6 years
  EQ-5D-5L is a validated questionnaire to assess the overall health-related quality of life in participants across diseases.
Parts 1 and 2: PROs in the European Organization for Research and Treatment of Cancer (EORTC) Quality of Life Questionnaire (QLQ-C30 [Core]) | Up to 6 years
  EORTC QLQ-C30 is validated questionnaire to assess overall health-related quality of life in participants with cancer.
Parts 1 and 2: PROs in the EORTC Quality of Life Questionnaire (Endometrial Cancer Module [QLQ-EN24]) | Up to 6 years
  EORTC QLQ-EN24 is a validated questionnaire to assess the overall health-related quality of life in participants with all stages of endometrial cancer.
Parts 1 and 2: Progression-free survival 2 (PFS2) | Up to 6 years
Parts 1 and 2: Number of participants with adverse events (AEs), Serious adverse events (SAEs) and treatment-emergent adverse events (TEAEs) | Up to 6 years
Parts 1 and 2: Number of participants with clinically significant changes in clinical laboratory parameters, physical examination, electrocardiogram (ECG) and participants reporting the intake of concomitant medication | Up to 6 years
Parts 1 and 2: Change from Baseline in vital sign: Diastolic Blood Pressure (DBP) and Systolic Blood Pressure (SBP) (Millimeters of mercury) | Baseline and up to 6 Years
Parts 1 and 2: Change from Baseline in vital sign: Heart Rate | Baseline and up to 6 Years
Parts 1 and 2: Change from Baseline in vital sign: Respiratory rate | Baseline and up to 6 Years
Parts 1 and 2: Change from Baseline in vital sign: Body temperature | Baseline and up to 6 Years
Parts 1 and 2: Number of participants with Eastern Cooperative Oncology Group (ECOG) Performance Status Scores | Up to 6 years
  Performance status will be assessed using the ECOG scale, with status score ranging from 0 to 5.
Parts 1 and 2: Minimum observed concentration (Cmin) and maximum observed concentration (Cmax) of dostarlimab (micrograms per milliliter) | Predose (Day 1) and postdose (Day 1) of Cycles 1, 2, 6, 7, 10, 15, and 20 (Cycle 1, 2, 6 is 21 days and Cycle 7, 10, 15, 20 is 42 days)
Parts 1 and 2: Cmin and Cmax at steady state of dostarlimab (micrograms per milliliter) | Predose (Day 1) and postdose (Day 1) of Cycles 1, 2, 6, 7, 10, 15, and 20 (Cycle 1, 2, 6 is 21 days and Cycle 7, 10, 15, 20 is 42 days)
Part 2: Cmin and Cmax of niraparib (nanograms per milliliter) | Predose (Day 1) and 3 hours postdose (Day 1) of Cycles 7 and 8 and Predose (Day 1) of Cycles 10 and 14 (each cycle is 42 days)
Part 2: Cmin and Cmax at steady state of niraparib (nanograms per milliliter) | Predose (Day 1) and 3 hours postdose (Day 1) of Cycles 7 and 8 and Predose (Day 1) of Cycles 10 and 14 (each cycle is 42 days)
Parts 1 and 2: Number of participants with anti-drug antibodies (ADA) against dostarlimab | Predose (Day 1)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (154):
- United States (52):
  - GSK Investigational Site, Phoenix, Arizona
  - GSK Investigational Site, Scottsdale, Arizona
  - GSK Investigational Site, Tucson, Arizona
  - GSK Investigational Site, Newport Beach, California
  - GSK Investigational Site, Palo Alto, California
  - GSK Investigational Site, Deerfield Beach, Florida
  - GSK Investigational Site, Jacksonville, Florida
  - GSK Investigational Site, Miami, Florida
  - GSK Investigational Site, Orlando, Florida
  - GSK Investigational Site, Atlanta, Georgia
  - GSK Investigational Site, Augusta, Georgia
  - GSK Investigational Site, Savannah, Georgia
  - GSK Investigational Site, Hinsdale, Illinois
  - GSK Investigational Site, Zion, Illinois
  - GSK Investigational Site, Fort Wayne, Indiana
  - GSK Investigational Site, Indianapolis, Indiana
  - GSK Investigational Site, Iowa City, Iowa
  - GSK Investigational Site, Lexington, Kentucky
  - GSK Investigational Site, Covington, Louisiana
  - GSK Investigational Site, New Orleans, Louisiana
  - GSK Investigational Site, Shreveport, Louisiana
  - GSK Investigational Site, Boston, Massachusetts
  - GSK Investigational Site, Springfield, Massachusetts
  - GSK Investigational Site, Detroit, Michigan
  - GSK Investigational Site, St Louis, Missouri
  - GSK Investigational Site, Lebanon, New Hampshire
  - GSK Investigational Site, Albuquerque, New Mexico
  - GSK Investigational Site, Rio Rancho, New Mexico
  - GSK Investigational Site, Albany, New York
  - GSK Investigational Site, Mineola, New York
  - GSK Investigational Site, New York, New York
  - GSK Investigational Site, The Bronx, New York
  - GSK Investigational Site, Charlotte, North Carolina
  - GSK Investigational Site, Durham, North Carolina
  - GSK Investigational Site, Kernersville, North Carolina
  - GSK Investigational Site, Mount Airy, North Carolina
  - GSK Investigational Site, Winston-Salem, North Carolina
  - GSK Investigational Site, Cincinnati, Ohio
  - GSK Investigational Site, Cleveland, Ohio
  - GSK Investigational Site, Columbus, Ohio
  - GSK Investigational Site, Hilliard, Ohio
  - GSK Investigational Site, Tulsa, Oklahoma
  - GSK Investigational Site, Philadelphia, Pennsylvania
  - GSK Investigational Site, Pittsburgh, Pennsylvania
  - GSK Investigational Site, Willow Grove, Pennsylvania
  - GSK Investigational Site, Providence, Rhode Island
  - GSK Investigational Site, Knoxville, Tennessee
  - GSK Investigational Site, Austin, Texas
  - GSK Investigational Site, Dallas, Texas
  - GSK Investigational Site, Charlottesville, Virginia
  - GSK Investigational Site, Roanoke, Virginia
  - GSK Investigational Site, Seattle, Washington
- Belarus (2):
  - GSK Investigational Site, Grodno
  - GSK Investigational Site, Minsk
- Belgium (3):
  - GSK Investigational Site, Aalst
  - GSK Investigational Site, Leuven
  - GSK Investigational Site, Liège
- Canada (7):
  - GSK Investigational Site, Calgary, Alberta
  - GSK Investigational Site, Winnipeg, Manitoba
  - GSK Investigational Site, Ottawa, Ontario
  - GSK Investigational Site, Sault Ste. Marie, Ontario
  - GSK Investigational Site, Toronto, Ontario
  - GSK Investigational Site, Montreal, Quebec
  - GSK Investigational Site, Québec, Quebec
- Czechia (2):
  - GSK Investigational Site, Brno
  - GSK Investigational Site, Prague
- Denmark (5):
  - GSK Investigational Site, Aalborg
  - GSK Investigational Site, Copenhagen
  - GSK Investigational Site, Herlev
  - GSK Investigational Site, Odense C
  - GSK Investigational Site, Roskilde
- Finland (3):
  - GSK Investigational Site, Kuopio
  - GSK Investigational Site, Tampere
  - GSK Investigational Site, Turku
- Germany (22):
  - GSK Investigational Site, Amberg
  - GSK Investigational Site, Bad Homburg
  - GSK Investigational Site, Cologne
  - GSK Investigational Site, Dessau
  - GSK Investigational Site, Dresden
  - GSK Investigational Site, Essen
  - GSK Investigational Site, Frankfurt
  - GSK Investigational Site, Giessen
  - GSK Investigational Site, Hamburg
  - GSK Investigational Site, Hanover
  - GSK Investigational Site, Jena
  - GSK Investigational Site, Karlsruhe
  - GSK Investigational Site, Kiel
  - GSK Investigational Site, Lübeck
  - GSK Investigational Site, Mainz
  - GSK Investigational Site, München
  - GSK Investigational Site, Offenbach
  - GSK Investigational Site, Ravensburg
  - GSK Investigational Site, Rosenheim
  - GSK Investigational Site, Tübingen
  - GSK Investigational Site, Ulm
  - GSK Investigational Site, Wiesbaden
- Greece (2):
  - GSK Investigational Site, Marousi
  - GSK Investigational Site, Thessaloniki
- Hungary (2):
  - GSK Investigational Site, Budapest
  - GSK Investigational Site, Debrecen
- Israel (7):
  - GSK Investigational Site, Ashkelon
  - GSK Investigational Site, Beersheba
  - GSK Investigational Site, Haifa
  - GSK Investigational Site, Jerusalem
  - GSK Investigational Site, Petah Tikva
  - GSK Investigational Site, Rehovot
  - GSK Investigational Site, Tel Aviv
- Italy (10):
  - GSK Investigational Site, Candiolo
  - GSK Investigational Site, Carpi MO
  - GSK Investigational Site, Lecce
  - GSK Investigational Site, Milan
  - GSK Investigational Site, Naples
  - GSK Investigational Site, Ponderano BI
  - GSK Investigational Site, Rome
  - GSK Investigational Site, Sassuolo
  - GSK Investigational Site, Trento
  - GSK Investigational Site, Udine
- Netherlands (6):
  - GSK Investigational Site, Amsterdam
  - GSK Investigational Site, Eindhoven
  - GSK Investigational Site, Enschede
  - GSK Investigational Site, Groningen
  - GSK Investigational Site, Maastricht
  - GSK Investigational Site, Rotterdam
- Norway (5):
  - GSK Investigational Site, Bergen
  - GSK Investigational Site, Oslo
  - GSK Investigational Site, Stavanger
  - GSK Investigational Site, Troms
  - GSK Investigational Site, Trondheim
- Poland (7):
  - GSK Investigational Site, Bialystok
  - GSK Investigational Site, Gdynia
  - GSK Investigational Site, Lodz
  - GSK Investigational Site, Olsztyn
  - GSK Investigational Site, Poznan
  - GSK Investigational Site, Szczecin
  - GSK Investigational Site, Warsaw
- Spain (6):
  - GSK Investigational Site, Barcelona
  - GSK Investigational Site, Donostia / San Sebastian
  - GSK Investigational Site, Madrid
  - GSK Investigational Site, Málaga
  - GSK Investigational Site, Murcia
  - GSK Investigational Site, Valencia
- Sweden (4):
  - GSK Investigational Site, Linköping
  - GSK Investigational Site, Lund
  - GSK Investigational Site, Stockholm
  - GSK Investigational Site, Uppsala
- Turkey (Türkiye) (3):
  - GSK Investigational Site, Adapazarı
  - GSK Investigational Site, Ankara
  - GSK Investigational Site, Istanbul
- Ukraine (2):
  - GSK Investigational Site, Chernihiv
  - GSK Investigational Site, Kharkiv
- United Kingdom (4):
  - GSK Investigational Site, Brighton
  - GSK Investigational Site, Cambridge
  - GSK Investigational Site, London
  - GSK Investigational Site, Truro

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to anonymized individual patient-level data (IPD) and related study documents of the eligible studies via the Data Sharing Portal. Details on GSK's data sharing criteria can be found at: https://www.gsk.com/en-gb/innovation/trials/data-transparency/
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Anonymized IPD will be made available within 6 months of publication of primary, key secondary and safety results for studies in product with approved indication(s) or terminated asset(s) across all indications.
Access Criteria: Anonymized IPD is shared with researchers whose proposals are approved by an Independent Review Panel and after a Data Sharing Agreement is in place. Access is provided for an initial period of 12 months but an extension may be granted, when justified, for up to 6 months.
URL: https://www.gsk.com/en-gb/innovation/trials/data-transparency/

REFERENCES:
- [Background] Mansoor R Mirza, Dana M Chase, Brian M Slomovitz, René dePont Christensen, Zoltán Novák, Destin Black, Lucy Gilbert, Sudarshan Sharma, Giorgio Valabrega, Lisa M Landrum, Lars C Hanker, Ashley Stuckey, Ingrid Boere, Michael A Gold, Annika Auranen, Bhavana Pothuri, David Cibula, Carolyn McCourt, Francesco Raspagliesi, Mark S Shahin, Sarah E Gill, Bradley J Monk, Joseph Buscema, Thomas J Herzog, Larry J Copeland, Min Tian, Zangdong He, Shadi Stevens, Eleftherios Zografos, Robert L Coleman, Matthew A Powell, . Dostarlimab for Primary Advanced or Recurrent Endometrial Cancer. The New England journal of medicine. 2023-Jun-08;388(23): 2145-2158. DOI : 10.1056/NEJMoa2216334 PMID: 36972026
- [Derived] Banerjee S, Ingles Russo Garces A, Garside J, Rahman T, Pearson C, Heffernan K. Real-world patient characteristics and survival outcomes in patients with advanced or recurrent endometrial cancer in England: a retrospective, population-based study. BMJ Open. 2024 Nov 24;14(11):e083540. doi: 10.1136/bmjopen-2023-083540. PMID 39581729
- [Derived] Auranen A, Powell MA, Sukhin V, Landrum LM, Ronzino G, Buscema J, Bauerschlag D, Lalisang R, Bender D, Gilbert L, Armstrong A, Safra T, Nevadunsky N, Sebastianelli A, Slomovitz B, Ring K, Coleman R, Podzielinski I, Stuckey A, Teneriello M, Gill S, Pothuri B, Willmott L, Sharma S, Dabrowski C, Antony G, Stevens S, Mirza MR, Fleming E. Safety of dostarlimab in combination with chemotherapy in patients with primary advanced or recurrent endometrial cancer in a phase III, randomized, placebo-controlled trial (ENGOT-EN6-NSGO/GOG-3031/RUBY). Ther Adv Med Oncol. 2024 Sep 28;16:17588359241277656. doi: 10.1177/17588359241277656. eCollection 2024. PMID 39346117
- [Derived] Valabrega G, Powell MA, Hietanen S, Miller EM, Novak Z, Holloway R, Denschlag D, Myers T, Thijs AM, Pennington KP, Gilbert L, Fleming E, Zub O, Landrum LM, Ataseven B, Gogoi R, Podzielinski I, Cloven N, Monk BJ, Sharma S, Herzog TJ, Stuckey A, Pothuri B, Secord AA, Chase D, Vincent V, Meyers O, Garside J, Mirza MR, Black D. Patient-reported outcomes in the subpopulation of patients with mismatch repair-deficient/microsatellite instability-high primary advanced or recurrent endometrial cancer treated with dostarlimab plus chemotherapy compared with chemotherapy alone in the ENGOT-EN6-NSGO/GOG3031/RUBY trial. Int J Gynecol Cancer. 2025 Jun;35(6):101852. doi: 10.1136/ijgc-2024-005484. Epub 2025 Apr 19. PMID 39322611
- [Derived] Mirza MR, Chase DM, Slomovitz BM, Christensen RD, Novak Z, Black D, Gilbert L, Sharma S, Valabrega G, Landrum LM, Hanker LC, Stuckey A, Boere I, Gold MA, Auranen A, Pothuri B, Cibula D, McCourt C, Raspagliesi F, Shahin MS, Gill SE, Monk BJ, Buscema J, Herzog TJ, Copeland LJ, Tian M, He Z, Stevens S, Zografos E, Coleman RL, Powell MA. A Plain Language Summary of "Dostarlimab for primary advanced or recurrent endometrial cancer". Future Oncol. 2025 Jan;21(2):151-168. doi: 10.2217/fon-2023-0940. Epub 2024 Jul 11. PMID 38990090
- [Derived] You M, Zeng X, Zhang J, Huang Y, Zhang Y, Cai Z, Hu Y. Cost-effectiveness analysis of dostarlimab plus carboplatin-paclitaxel as first-line treatment for advanced endometrial cancer. Front Immunol. 2023 Sep 4;14:1267322. doi: 10.3389/fimmu.2023.1267322. eCollection 2023. PMID 37731489
- [Derived] Morton M, Marcu I, Levine M, Cosgrove C, Backes F, O'Malley D, Chambers L. Evaluation of Efficacy and Adverse Events After Second Immunotherapy Exposure in Endometrial and Cervical Carcinoma. Obstet Gynecol. 2023 Aug 1;142(2):360-363. doi: 10.1097/AOG.0000000000005243. Epub 2023 Jul 5. PMID 37411031
- [Derived] Mirza MR, Chase DM, Slomovitz BM, dePont Christensen R, Novak Z, Black D, Gilbert L, Sharma S, Valabrega G, Landrum LM, Hanker LC, Stuckey A, Boere I, Gold MA, Auranen A, Pothuri B, Cibula D, McCourt C, Raspagliesi F, Shahin MS, Gill SE, Monk BJ, Buscema J, Herzog TJ, Copeland LJ, Tian M, He Z, Stevens S, Zografos E, Coleman RL, Powell MA; RUBY Investigators. Dostarlimab for Primary Advanced or Recurrent Endometrial Cancer. N Engl J Med. 2023 Jun 8;388(23):2145-2158. doi: 10.1056/NEJMoa2216334. Epub 2023 Mar 27. PMID 36972026